CLINICAL TRIAL: NCT06660875
Title: Comparison of Postoperative Analgesic Efficacy of Serratus Posterior Superıor Intercostal Plane Block and Combination of Interscalene Brachial Plexus Block and Superfisial Plexus Block in Shoulder Arthroscopies
Brief Title: Comparison of Postoperative Analgesic Efficacy of SPSIPB and Combination of IBPB and SCPB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Muruvvet Taskir Turan, Principal investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AEŞH-BADEK-1003-2024
Record Dates: First submitted 2024-10-11; First posted 2024-10-28 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Shoulder Arthroscopy; İnterscalene Brachial Plexus Block; Superficial Cervical Plexus Block; Serratus Posterior Superior Intercostal Plane Block
Keywords: Remifantanile conception; Acute pain; Postoperatif pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus posterior superior intercostal plane block (Active Comparator): With the patient in the prone position the skin is disinfected .Linear USG probe is placed on the spine of the scapula using an in-plane technique and moved medially. The 3rd rib is identified just on the medial scapular border. After visualizing the trapezius, rhomboid major, and serratus posterior superior muscles (from top to bottom) under USG guidance, a 22-G X 80-mm block needle is directed caudally and advanced until it contacted the rib. To confirm and obtain a plane between the serratus posterior superior and intercostal muscles, hydrodissection is performed using 2 ml of isotonic solution. After the needle site is confirmed, 30 ml of 0.25% bupivacaine is injected ; the local anesthetic spread is confirmed by USG.
  Interventions: Drug: Serratus posterior superior intercostal plane block
- Interscalene brachial plexus block and superficial cervical plexus block (Active Comparator): İBPB:While the patient is in the supine position, the ultrasound probe is placed on the cricoid cartilage and moved laterally to visualize the trachea, thyroid, carotid artery, internal jugular vein, and sternocleidomastoid muscle. The brachial plexus is identified by directing it posteriorly and laterally between the anterior and middle scalene muscles. After entering between the roots using the in-plane technique and confirming the location with a 2 ml isotonic sodium injection, 20 ml of 0.25% bupivacaine is injected.
  SCPB:While the patient is in the supine position, the ultrasound probe is placed at the midpoint of the sternocleidomastoid (SCM) muscle. The cervical plexus is visualized deep to the posterior border of the SCM muscle. The needle is inserted deep to the SCM, directed towards the levator scapula. After confirming the location with a 2 ml isotonic sodium injection, 10 ml of 0.25% bupivacaine is injected.
  Interventions: Drug: Interscalene brachial plexus block and superficial cervical plexus block

INTERVENTIONS:
Drug: Serratus posterior superior intercostal plane block — Serratus posterior superior intercostal plane block is performed, under US guidance, before the surgical operation, and the induction of anesthesia, and when the patient is placed in the prone position.
  Arms: Serratus posterior superior intercostal plane block
Drug: Interscalene brachial plexus block and superficial cervical plexus block — İnterscalene brachial plexus block and superficial cervical plexus block is performed, under US guidance, before the surgical operation, and the induction of anesthesia, and when the patient is placed in the prone position.
  Arms: Interscalene brachial plexus block and superficial cervical plexus block

SUMMARY:
Shoulder arthroscopy is one of the frequently performed surgical procedures today. After shoulder surgery, ensuring sufficent analgesia is necessary for both the patient's comfort and for the early and regular performance of the required postoperative rehabilitation exercises. Nerve blocks provide better pain control, opioid consumption in the postoperative period, and consequently have advantages such as fewer side effects and lower risks of pulmonary and cardiac complications. Multimodal analgesia approach is preferred for patients undergoing shoulder arthroscopy. Along with intravenous analgesic agents, peripheral nerve blocks (applied to every suitable and consenting patient) are performed based on patient preference. This study aims to compare the analgesic efficacy in the postoperative period of patients undergoing shoulder arthroscopy with a combination of interscalene brachial plexus block and superficial cervical plexus block with serratus posterior superior intercostal plane block.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* American Society of Anesthesiologists (ASA) physical status I-II-III
* Body mass index 18 to 30 kg/m2
* Elective shoulder arthroscopy surgery

Exclusion Criteria:

* Under 18 and over 65
* ASA score IV and above
* Advanced co-morbidity
* History of bleeding diathesis
* BMI under 18 kg/m2 and over 30 kg/m2
* Patient refusing the procedure
* Patients who have previously undergone shoulder surgery
* Chronic opioid or analgesic use
* Patients who will operate under emergency conditions
* Patients who will not undergo shoulder surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-10-11 (Estimated); Study Completion 2025-10-21 (Estimated)

PRIMARY OUTCOMES:
Intraoperative remifentanil consumption | During The intraoperatif period
  The amount of remifentanil that patients need to maintain anesthesia during the intraoperative period will be recorded

SECONDARY OUTCOMES:
Pain scores | First 24 hours after surgery
  Pain will be assessed at rest and while movement using the from 0 (no pain) to 10 (worst pain). Pain assessment will be done at the 1st, 2nd, 4th, 12th, and 24th hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Yenimahalle, Ankara, Turkey (Türkiye)